CLINICAL TRIAL: NCT00685828
Title: Phase III Randomized, Intergroup, International Trial Assessing the Clinical Activity of STI-571 at Two Dose Levels in Patients With Unresectable or Metastatic Gastrointestinal Stromal Tumors (GIST) Expressing the KIT Receptor Tyrosine Kinase (CD117)
Brief Title: Imatinib Mesylate in Treating Patients With Unresectable or Metastatic Gastrointestinal Stromal Tumor
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Italian Sarcoma Group (Network); Australasian Gastro-Intestinal Trials Group (Network); Scandinavian Sarcoma Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-62005; EORTC-62005; AGITG-AGO102-GIST; ISG-62005; SSG-15
Record Dates: First submitted 2008-05-22; First posted 2008-05-28 (Estimated); Last update posted 2014-07-04 (Estimated); Status verified 2014-07

CONDITIONS: Gastrointestinal Stromal Tumor
Keywords: gastrointestinal stromal tumor
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — Imatinib Mesylate

ARMS (2):
- Arm I (Active Comparator): Patients receive low-dose oral imatinib mesylate once daily in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: imatinib mesylate
- Arm II (Experimental): Patients receive high-dose oral imatinib mesylate twice daily in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: imatinib mesylate

INTERVENTIONS:
Drug: imatinib mesylate — By mouth

SUMMARY:
RATIONALE: Imatinib mesylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known which dose of imatinib mesylate is more effective in treating gastrointestinal stromal tumor.

PURPOSE: This randomized phase III trial is studying two different doses of imatinib mesylate to compare how well they work in treating patients with unresectable or metastatic gastrointestinal stromal tumor.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare outcomes of patients with unresectable or metastatic gastrointestinal stromal tumor that expresses KIT (CD117) treated with low-dose imatinib mesylate vs high-dose imatinib mesylate.

Secondary

* To assess response rates in patients treated with two different doses of imatinib mesylate.
* To assess the toxicities of two different doses of imatinib mesylate in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to participating center, measurability of disease (measurable vs non-measurable), and WHO performance status (0-2 vs 3). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive low-dose oral imatinib mesylate once daily in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive high-dose oral imatinib mesylate twice daily in the absence of disease progression or unacceptable toxicity.

In the event of disease progression, patients on arm I may cross over to arm II and receive high-dose imatinib mesylate. Patients who continue to progress despite treatment with high-dose imatinib mesylate are removed from the study.

After completion of study therapy, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed gastrointestinal stromal tumor (GIST)

  * Metastatic or unresectable disease
* Immunohistochemical confirmation of KIT (CD117) expression by tumor as documented by DAKO antibody staining
* Measurable or non-measurable disease by conventional imaging (CT scan or MRI) or physical examination

  * If a target lesion has been previously embolized or irradiated, there must be objective evidence of progression to be considered for response assessment
* No known brain metastasis

PATIENT CHARACTERISTICS:

* WHO performance status 0-3
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN (≤ 5 times ULN if hepatic metastases are present)
* Creatinine ≤ 1.5 times ULN
* ANC ≥ 1,000/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9 g/dL (transfusions allowed)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for up to 3 months after completion of study therapy
* No NYHA class III-IV cardiac disease
* No congestive heart failure or myocardial infarction within the past 2 months
* No severe and/or uncontrolled concurrent medical disease (e.g., uncontrolled diabetes, uncontrolled chronic renal or liver disease, or active uncontrolled infection [e.g., HIV])
* No other prior malignancy except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for 5 years
* No medical, psychological, familial, sociological, or geographical condition that, in the opinion of the investigator, may preclude the patient's ability to tolerate or complete study treatment, comply with study protocol and follow-up schedule, or give reliable informed consent

PRIOR CONCURRENT THERAPY:

* Recovered from all prior therapy
* More than 28 days since prior chemotherapy, biologic therapy, or any other investigational drug
* More than 14 days since prior major surgery
* No concurrent therapeutic anticoagulation with coumarin derivatives

  * Concurrent therapeutic anticoagulation with low-molecular weight heparin allowed
  * Concurrent mini-dose coumarin derivatives (i.e., equivalent to 1 mg of oral warfarin daily) as prophylaxis allowed
* No concurrent cytokines (i.e., filgrastim [G-CSF] or sargramostim [GM-CSF]) to support blood counts
* No other concurrent investigational drugs
* No other concurrent anticancer agents, including chemotherapy, radiotherapy, or anticancer biologic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 946 (Actual)
Dates: Start 2001-01; Primary Completion 2002-02 (Actual)

PRIMARY OUTCOMES:
Progression-free survival

SECONDARY OUTCOMES:
Overall survival
Objective tumor response
Toxicity as assessed by NCI CTC v2.0

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Verweij, MD, PhD, Study Chair — Daniel Den Hoed Cancer Center at Erasmus Medical Center; Paolo G. Casali, MD, Study Chair — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano; John R. Zalcberg, MB, BS, PhD, FRACP, Study Chair — Peter MacCallum Cancer Centre, Australia; Kirsten Sundby Hall, MD, Study Chair — Lund University Hospital

REFERENCES:
- [Background] Judson I. Imatinib in advanced gastrointestinal stromal tumour: when is 800 mg the correct dose? Curr Opin Oncol. 2008 Jul;20(4):433-7. doi: 10.1097/CCO.0b013e328302ed96. PMID 18525340
- [Background] van Glabbeke MM, Owzar K, Rankin C, et al.: Comparison of two doses of imatinib for the treatment of unresectable or metastatic gastrointestinal stromal tumors (GIST): a meta-analyis based on 1,640 patients (pts). [Abstract] J Clin Oncol 25 (Suppl 18): A-10004, 546s, 2007.
- [Result] Le Cesne A, Van Glabbeke M, Verweij J, Casali PG, Findlay M, Reichardt P, Issels R, Judson I, Schoffski P, Leyvraz S, Bui B, Hogendoorn PC, Sciot R, Blay JY. Absence of progression as assessed by response evaluation criteria in solid tumors predicts survival in advanced GI stromal tumors treated with imatinib mesylate: the intergroup EORTC-ISG-AGITG phase III trial. J Clin Oncol. 2009 Aug 20;27(24):3969-74. doi: 10.1200/JCO.2008.21.3330. Epub 2009 Jul 20. PMID 19620483
- [Result] Van Glabbeke MM, Verweij J, Casali P, et al.: Type of progression in patients treated with imatinib for advanced gastrointestinal stromal tumor (GIST): A study based on the EORTC-ISG-AGITG trial 62005. [Abstract] J Clin Oncol 27 (Suppl 15): A-10536, 2009.
- [Result] Sciot R, Debiec-Rychter M, Daugaard S, Fisher C, Collin F, van Glabbeke M, Verweij J, Blay JY, Hogendoorn PC; EORTC Soft Tissue and Bone Sarcoma Group; Italian Sarcoma Group; Australasian Trials Group. Distribution and prognostic value of histopathologic data and immunohistochemical markers in gastrointestinal stromal tumours (GISTs): An analysis of the EORTC phase III trial of treatment of metastatic GISTs with imatinib mesylate. Eur J Cancer. 2008 Sep;44(13):1855-60. doi: 10.1016/j.ejca.2008.06.003. Epub 2008 Jul 22. PMID 18653326
- [Result] Verweij J, Casali PG, Kotasek D, Le Cesne A, Reichard P, Judson IR, Issels R, van Oosterom AT, Van Glabbeke M, Blay JY. Imatinib does not induce cardiac left ventricular failure in gastrointestinal stromal tumours patients: analysis of EORTC-ISG-AGITG study 62005. Eur J Cancer. 2007 Apr;43(6):974-8. doi: 10.1016/j.ejca.2007.01.018. Epub 2007 Mar 2. PMID 17336514
- [Result] Debiec-Rychter M, Sciot R, Le Cesne A, Schlemmer M, Hohenberger P, van Oosterom AT, Blay JY, Leyvraz S, Stul M, Casali PG, Zalcberg J, Verweij J, Van Glabbeke M, Hagemeijer A, Judson I; EORTC Soft Tissue and Bone Sarcoma Group; Italian Sarcoma Group; Australasian GastroIntestinal Trials Group. KIT mutations and dose selection for imatinib in patients with advanced gastrointestinal stromal tumours. Eur J Cancer. 2006 May;42(8):1093-103. doi: 10.1016/j.ejca.2006.01.030. Epub 2006 Apr 18. PMID 16624552
- [Result] Van Glabbeke M, Verweij J, Casali PG, Simes J, Le Cesne A, Reichardt P, Issels R, Judson IR, van Oosterom AT, Blay JY. Predicting toxicities for patients with advanced gastrointestinal stromal tumours treated with imatinib: a study of the European Organisation for Research and Treatment of Cancer, the Italian Sarcoma Group, and the Australasian Gastro-Intestinal Trials Group (EORTC-ISG-AGITG). Eur J Cancer. 2006 Sep;42(14):2277-85. doi: 10.1016/j.ejca.2006.03.029. Epub 2006 Jul 28. PMID 16876399
- [Result] Van Glabbeke M, Verweij J, Casali PG, Le Cesne A, Hohenberger P, Ray-Coquard I, Schlemmer M, van Oosterom AT, Goldstein D, Sciot R, Hogendoorn PC, Brown M, Bertulli R, Judson IR. Initial and late resistance to imatinib in advanced gastrointestinal stromal tumors are predicted by different prognostic factors: a European Organisation for Research and Treatment of Cancer-Italian Sarcoma Group-Australasian Gastrointestinal Trials Group study. J Clin Oncol. 2005 Aug 20;23(24):5795-804. doi: 10.1200/JCO.2005.11.601. PMID 16110036
- [Result] Verweij J, Casali PG, Zalcberg J, et al.: Early efficacy comparison of two doses of imatinib for the treatment of advanced gastro-intestinal stromal tumors (GIST): interim results of a randomized phase III trial from the EORTC-STBSG, ISG and AGITG. [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-3272, 814, 2003.